CLINICAL TRIAL: NCT06661616
Title: Cognitive Effects Associated With Hippocampal Neurogenesis Induced by Electroconvulsive Therapy in the Treatment of Depression
Brief Title: Cognitive Effects Associated With Hippocampal Neurogenesis Induced by ECT in the Treatment of Depression
Acronym: CONHECT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D17-P018
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder (MDD); Bipolar Disorder Depression
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of blood plasma and peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Depressed patient treated with electroconvulsivotherapy: The indication for ECT treatment is established by the department's medical team. Participants are not assigned to ECT as part of this observational study.
- Depressed patient treated without electroconvulsivotherapy: The indication for antidepressant treatment is established by the department's medical team. Participants are not assigned to ECT as part of this observational study.
- Healthy volunteers: Age- and sex-matched healthy volunteers free of psychiatric disorders.

SUMMARY:
Electroconvulsive therapy (ECT) is the treatment of choice for drug-resistant depression (30% of patients), or when there is a short-term risk to the patient's life. Despite its robust efficacy and rapid onset of action, its use is limited both by the limited range of treatment available and by the cognitive effects sometimes induced. The present study focuses on the links between the efficacy of ECT, its cognitive effects and the formation of new neurons in the hippocampus (hippocampal neurogenesis) associated with this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Study population: depressed subjects treated with ECT

   * Male or female over 18 years of age
   * Hospitalised at the Centre Hospitalier Sainte-Anne
   * Suffering from a unipolar or bipolar major depressive episode, according to DSM5 criteria
   * Indication for ECT treatment
   * Patient has given informed written consent
   * Beneficiary of a social security scheme
2. Control population: depressed subjects treated without ECT

   * Male or female over 18 years of age
   * Hospitalised at the Centre Hospitalier Sainte-Anne
   * Suffering from a unipolar or bipolar major depressive episode, according to DSM5 criteria
   * Patient who has given informed written consent
   * Beneficiary of a social security scheme
3. Control population: healthy volunteers

   * Male or female over 18 years of age
   * Patient with written informed consent
   * Beneficiary of a social security scheme

Exclusion Criteria:

1. Study population: depressed subjects with ECT

   * Psychiatric comorbidity: schizophrenia, pervasive developmental disorder, dependence on a substance other than tobacco
   * Neurological comorbidity: Parkinson's disease, dementia
   * ECT treatment in the 6 months prior to inclusion
   * Compulsory care
   * Protected adults, persons under court protection measures
   * Persons deprived of liberty by judicial or administrative decision;
   * Refusal of consent to ECT treatment
   * Contraindications to ECT (HTIC, recent history of stroke, severe uncontrolled arterial hypertension, contraindication to anaesthesia)
   * Contraindications to MRI (patients with metal prostheses, claustrophobia)
   * Pregnant or breast-feeding women
2. Control population: depressed subjects without ECT

   * Psychiatric comorbidity: schizophrenia, pervasive developmental disorder, dependence on any substance other than tobacco
   * Neurological comorbidity: Parkinson's disease, dementia
   * ECT treatment in the 6 months prior to inclusion
   * Compulsory care
   * Protected adults, persons under court protection measures
   * Persons deprived of liberty by judicial or administrative decision;
   * Pregnant or breast-feeding women
3. Control population: healthyvolunteers

   * Protected adults, persons under legal protection,
   * Persons deprived of their liberty by judicial or administrative decision ;
   * persons hospitalised for purposes other than research
   * Clear psychiatric history
   * Dependence on any substance other than tobacco
   * Neurological history: Parkinson's disease, dementia
   * Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study focuses on a population of adult patients suffering from unipolar or bipolar depression and treated with electroconvulsive therapy.
  In order to monitor the impact of depression on cognitive functions, including memory, and on biological markers and brain imaging, 35 depressed subjects treated without ECT will be recruited.
  And to monitor the effect of time on memory, 35 healthy volunteers will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Correlation between increased hippocampal volume and post-ECT retrograde amnesia | After a course of ECT, up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Anne Hospital (GHU Paris Psychiatrie et Neurosciences), Paris, France